CLINICAL TRIAL: NCT02348853
Title: Intervention for Sustainable Weight Loss in Military Families
Brief Title: Healthy Families Healthy Forces Study
Acronym: HF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Roberts, Senior Scientist & Director, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13035001
Record Dates: First submitted 2015-01-13; First posted 2015-01-28 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Weight For Living (HWL) (Experimental): HWL is a behavioral intervention designed to effectively facilitate hunger suppression with several concurrent approaches. Hunger suppression is a core behavioral goal of the intervention, and strategies will be used to support that goal, for example increasing meal frequency and encouraging the use of highly satiating low-energy foods to reduce hunger acutely. A unique combination of healthy dietary goals will be recommended that support hunger suppression and/or maintenance of satiety: high total dietary fiber, moderately high protein, moderately low glycemic load (GL) and low energy density.
  Interventions: Behavioral: Healthy Weight for Living (HWL)
- Current Best Practice (CBP) (Experimental): This intervention is an adapted version of Group Lifestyle Balance which is a validated weight loss program for community groups and military populations that is an official adaptation of the gold standard Diabetes Prevention Program Lifestyle Balance intensive research intervention. It has both training programs for interventionists and program material available on the web and is also slightly modified from the Diabetes Prevention Program study to take into account changing national nutrition recommendations.
  Interventions: Behavioral: Current Best Practice (CBP)

INTERVENTIONS:
Behavioral: Healthy Weight for Living (HWL)
  Arms: Healthy Weight For Living (HWL)
Behavioral: Current Best Practice (CBP)
  Arms: Current Best Practice (CBP)

SUMMARY:
U.S. Army Medical Research & Materiel Command Telemedicine and Advanced Technology Research Center (TATRC) is sponsoring the HF2 (Healthy Families, Healthy Forces) Study. This is a randomized trial comparing two different interventions for sustainable weight loss. Specifically, the investigators will compare a "current best practice (CBP)" intervention that includes standard dietary advice with a new, "Healthy Weight for Living (HWL)" intervention that includes recommendations to eat a diet rich in protein, dietary fiber, low glycemic index carbohydrates and low calorie foods. The objective of this study is to compare the CBP and HWL interventions when delivered to adult dependents of active duty (AD) military personnel and measure weight loss effects in both the adult dependents and the AD military personnel they live with.

DETAILED DESCRIPTION:
This is a randomized trial comparing two different interventions for sustainable weight loss. Specifically researchers will compare a current best practice (CBP) intervention that includes standard dietary advice with a new Healthy Weight for Living (HWL) intervention that includes recommendations to eat a diet rich in protein, dietary fiber and low glycemic index carbohydrates. The population will be adult dependents of Active Duty (AD) military personnel or retired military personnel (direct intervention participants) and the AD or retired military personnel they live with (indirect intervention participants). The primary outcome will be weight change from baseline to 1 year in the adult dependents. The objective of this study is to compare the CBP and HWL interventions when delivered to adult dependents of AD or retired military personnel and measure weight loss effects in both the adult dependents and the AD or retired military personnel they live with. The working hypothesis is that that the HWL intervention will result in significantly greater weight loss over 1 year than the CBP intervention in an intent-to-treat analysis in adult dependents, and that the greater weight loss in HWL will be associated with greater management of hunger and greater adherence to the goal of reducing energy intake. Weight change up until the 18-24 month period will be measured as a secondary outcome in a cohort of participants who will reach the 18-24 month milestone in the study on or prior to December, 2018. A per protocol analysis will also be applied for comparison of the two weight loss arms. (In addition, weight change will be measured in the participants' AD or retired military personnel partner to test the hypothesis that there is a ripple effect of benefits from the interventions associated with effects in the primary recipients.) The original study plan was to examine weight change over 2 years but due to slower recruiting than anticipated the hypotheses were revised to allow for 1 year to be the primary outcome, with secondary outcomes in the subgroup followed until 18-24 months.

The researchers plan to test our central hypothesis and accomplish the study objectives with the following technical objectives:

1. Conduct a randomized trial comparing the HWL intervention to the CBP intervention over 1 year in adult dependents of AD or retired military personnel. The primary outcome will be weight change from baseline to 1 year. The working hypothesis is that randomization to the HWL intervention will result in significantly greater weight loss over 1 year than randomization to the CBP intervention, and that greater weight loss in the HWL intervention will be associated with greater adherence to the goals of reducing energy intake and hunger.
2. Compare the change in weight loss of participants in the HWL intervention to the CBP intervention over the 18-24 month timepoints in the subgroup of participants who will reach the 18-24 month milestone on or prior to December, 2018. The working hypothesis is that randomization to the HWL intervention will result in significantly improved weight loss retention compared to randomization to the CBP intervention.
3. Examine the effects of the interventions delivered to adult dependents of AD or retired military personnel on the weight of AD or retired military personnel themselves. The working hypothesis, based on preliminary data, is that there will be a "ripple" effect of program benefits from intervention participants to the AD or retired military personnel they live with; specifically, overweight and obese AD or retired military personnel will lose more weight if their partner is randomized to the HWL intervention compared to the CBP intervention, because the weight loss of AD or retired military personnel indirectly exposed to the intervention will be proportional to the weight loss of their adult dependent who is directly exposed.
4. Compare the effects of the two interventions on changes in cardiometabolic risk factors. The working hypothesis is that there will be significantly greater improvements between baseline and 1 year in key cardiometabolic risk factors in adult dependents enrolled in the HWL intervention compared to the CBP intervention, and differences between groups will be predicted by differences in weight loss. For a select subgroup of participants who reach the 18-24 month timepoint on or prior to December 2018, the working hypothesis is that there will be significantly greater improvements in between baseline and 2 years in key cardiometabolic risk factors in adult dependents enrolled in the HWL compared to the CBP intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult dependent of active duty (AD) military personnel: an individual who is at least 18 years and have a military identification(ID) card indicating they are a dependent.
* This includes AD military sponsor's children at least 18 years of age (by birth or adoption), spouse, partner, parents, and parent-in-laws)
* At the time of enrollment, willing to be randomized to one of the intervention groups and complete outcome assessments, at least 18 years old at time of provision of informed consent
* BMI at screening greater than or equal to 25.0 kg/m2
* English speaking
* AD military personnel: AD military personnel do not have to meet any criteria other than having an adult partner enrolled in the weight loss program.

Exclusion Criteria:

* Adult dependent of AD military personnel: BMI <25
* Pregnant
* Expecting to become pregnant within duration of the study, or lactating
* Prior weight loss surgery
* Concurrent participation in another weight loss program or research study
* Non-English speaking
* Currently undergoing divorce proceedings
* Very active individuals (> 2 hours/day vigorous activity)
* Individuals who have lost > 10 lb in the past 6 months
* Individuals with thyroid disease who have had changes in medications within the past 3 months
* Individuals with Type 1 diabetes and individuals with Type 2 diabetes who started using insulin in childhood (before 18 years)
* Those with stomach or intestinal resection, including gastric bypass or other weight loss surgery that influences food intake or absorption of food
* Those with eating disorder such as anorexia, bulimia or binge-eating disorder currently or within the past 5 years
* Those with diagnosis of celiac disease, inflammatory bowel disease or any condition that influences ability to absorb food
* Those with current moderate to severe depression that prevents individual engaging in work or usual activities
* Those with recent unstable heart disease, myocardial infarction
* Active cancer
* Taking medication for severe kidney disease
* Chronic obstructive pulmonary disease
* Immunologic disorders
* AIDS
* Schizophrenia
* Psychosis or bipolar disorder
* Individuals who drink >3 drinks daily or >20 drinks/week
* Individuals with other diseases or taking other medications that impact ability to comply with the intervention core goal of achieving weight loss of 1-2 lb per week through some combination of changing types and amounts of consumed foods and exercise
* Excluded medications include steroids except topical preparations.
* AD military personnel: Those not currently living with the dependent due to separation and/or divorce proceedings will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Weight change in adult dependents of active duty military | Baseline to 12 months
  weight change from baseline to 12 months

SECONDARY OUTCOMES:
change in systolic and diastolic blood pressure (mmHg) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
change in total cholesterol (mg/dL) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
change in HDL cholesterol (mg/dL) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
change in LDL cholesterol (mg/dL) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
change in triacylglycerol (mg/dL) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
change in serum glucose (mg/dL) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
change in serum insulin (μIU/mL) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
change in homeostasis model assessment-estimated insulin resistance (HOMA-IR) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
change in C-reactive protein (CRP) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
change in HbA1c | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
emotional eating as measured by the Three Factor Eating Questionnaire - r18 (TFEQ-r18) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  TFEQ-r18 measures the cognitive and behavioral aspects of eating and has three subscales: cognitive restraint (CR), uncontrolled eating (UE), and emotional eating (EE). The score range for EE is 3 - 12, and higher scores indicate greater emotional eating. The EE subscale has 3 items, each on a 4-point Likert scale (1 - 4). The items are summed up for each subscale, and the total CR, UE, and EE scores are considered separately.
food cravings as measured by the Food Craving Questionnaire (FCQ) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  Food Cravings Questionnaire - State (FCQ-S) measures situational food cravings. It has 15 items, each of which is on a 5-point Likert scale (1 - 5), and the score range is 15 - 75. Higher scores indicate situational food cravings of greater intensity. Scores on all items are summed up for a total score.
  Food Cravings Questionnaire - Trait (FCQ-T) measures frequency and intensity of food cravings. It has 39 items, each of which is on a 6-point Likert scale (1 - 6), and the score range is 39 - 234. Higher scores indicate more frequent and intense food cravings. Scores on all items are summed up for a total score.
dietary intake as measured by 24-hour recalls and supermarket receipts | baseline to 6 months, 12 months, and 18/24 months
uncontrolled eating as measured by the Three Factor Eating Questionnaire - r18 (TFEQ-r18) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  TFEQ-r18 measures the cognitive and behavioral aspects of eating and has three subscales: cognitive restraint (CR), uncontrolled eating (UE), and emotional eating (EE). The score range for UE is 9 - 36, and higher scores indicate greater uncontrolled eating. The UE subscale has 9 items, each on a 4-point Likert scale (1 - 4). The items are summed up for each subscale, and the total CR, UE, and EE scores are considered separately.
cognitive restraint as measured by the Three Factor Eating Questionnaire - r18 (TFEQ-r18) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  TFEQ-r18 measures the cognitive and behavioral aspects of eating and has three subscales: cognitive restraint (CR), uncontrolled eating (UE), and emotional eating (EE). The score range for CR is 6 - 24, and higher scores indicate greater cognitive restraint. The CR subscale has 6 items, each on a 4-point Likert scale (1 - 4). The items are summed up for each subscale, and the total CR, UE, and EE scores are considered separately.
Weight change in adult dependents of active duty military, 18-24 months | baseline to 18 months, 24 months
  Weight change up until the 18-24 month period will be measured in a cohort of participants who will reach the 18-24 month milestone in the study on or prior to December, 2018
weight change in active duty military | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months

OTHER OUTCOMES:
physical activity as measured by the 7-Day Stanford Physical Activity Recall | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  The 7-Day Stanford Physical Activity Recall estimates an individual's time spent in sleep and physical activity for the 7 days prior to the interview. Energy expenditure based on time spent in sleep and physical activities can be estimated. Sub-scores of energy expenditure for each of the following activities are calculated, summed, and averaged to estimate energy expenditure as kilocalories per day: sleep, moderate physical activity, hard physical activity, and very hard physical activity. Higher scores indicate greater physical activity per day. Metabolic equivalent (MET) value for each activity is provided: 1 MET for sleep, 4 METs for moderate activity, 6 METs for hard activity, and 10 METs for very hard activity. Time spent in each activity over 7 days is multiplied by the appropriate MET value. Plausible minimum and maximum values are not provided.
quality of life as measured by the RAND 36-Item Health Survey, Short Form (SF-36) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  SF-36 measures eight aspects of health: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Perceived change in health is also assessed. Each of the subscales (8 aspects of health and perceived change) has a score range of 0 - 100. The composite score also has a score range of 0 - 100. Higher scores indicate more favorable health states. Each item is on a Likert scale, which is either 3 points (1 - 3) or 5 points (1 - 5). The protocol provides a transformed score for response to each item, and the transformed scores of the 9 subscales are averaged to derive a composite score between 0 and 100.
Duke Social Support and Stress Scale (DUSOCS) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  The DUSOCS measures perceived levels of social support and stress experienced from family and non-family social ties. There are six subscales: Family Support, Non-Family Support, Social Support (composite of Family and Non-Family Support), Family Stress, Non-Family Stress, and Social Stress (composite of Family and Non-Family Stress). The score range is 0 - 100 for each subscale. Higher scores on the Support and Stress scales indicate higher levels of perceived social support and stress, respectively. For each subscale, responses are summed up as raw scores. The raw scores are divided by the appropriate factors and multiplied by 100, resulting in a scaled score between 0 and 100. Calculation for Social Support involves summing up items related to Family Support and Non-Family Support and hence provides a composite score for the two sources of social support. Similarly, calculation for Social Stress involves summing up items related to Family Stress and Non-Family Stress.
Perceived Stress Scale (PSS) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  The PSS measures how different situations can affect emotions and perceived stress. The score range is 0 - 40. Higher scores indicate higher levels of perceived stress. There are 10 items, each of which is on a 5-point Likert scale (0 - 4). Four of the items require reverse coding. The score is determined by summing up responses to the 10 items.
Pittsburgh Sleep Quality Index (PSQI) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  The PSQI measures sleep quality and disturbance over the course of one month. There are seven subscales: subjective sleep quality, sleep latency, sleep duration, 4. habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The scoring range of each subscale is 0 - 3. The scoring range of the Global PSQI (the composite score of the seven subscales) is 0 - 21. For both the subscales and Global PSQI, higher scores indicate greater difficulties with sleeping. Subscales 1, 3, and 6 each consist of only one item, and no scoring calculations are applied. Subscales 2, 5, and 7 have multiple items that are summed up as raw scores, and the protocol provides the corresponding transformed scores. Subscale 4 calculates habitual sleep efficiency (Number of hours slept/Number of hours spent in bed x 100%) and assigns a transformed score. Global PSQI is the sum of the seven transformed scores.
World Health Organization Quality of Life, Short Form (WHOQOL-BREF) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  The WHOQOL-BREF measures four domains of health: physical health, psychological health, social relationships, and environment. Each measured domain has a score range of 0 - 100. Higher scores indicate higher quality of life with respect to each domain of health. There are 26 items, 24 of which are used for calculations (7 items for physical health, 6 items for psychological health, 3 items for social relationships, and 8 items for environment). Each item is on a 5-point Likert scale (1 - 5), and three negatively phrased items require reverse coding. The point values are summed up as raw scores, and the protocol provides the transformed score for each raw score.
Beck Depression Inventory (BDI-II) | baseline to 6 months, 12 months, 24 months and 12 months - 18/24 months
  The BDI-II measures depression severity. The score range is 0 - 63, and higher scores indicate greater depression severity. Nineteen items are on a 4-point Likert scale (0 - 3). Two items are on a 7-point Likert scale, and responses are scaled to 0 - 3. The values are summed up to calculate the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Roberts, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Das SK, Bukhari AS, Taetzsch AG, Ernst AK, Rogers GT, Gilhooly CH, Hatch-McChesney A, Blanchard CM, Livingston KA, Silver RE, Martin E, McGraw SM, Chin MK, Vail TA, Lutz LJ, Montain SJ, Pittas AG, Lichtenstein AH, Allison DB, Dickinson S, Chen X, Saltzman E, Young AJ, Roberts SB. Randomized trial of a novel lifestyle intervention compared with the Diabetes Prevention Program for weight loss in adult dependents of military service members. Am J Clin Nutr. 2021 Oct 4;114(4):1546-1559. doi: 10.1093/ajcn/nqab259. PMID 34375387

DOCUMENTS (1):
  • Informed Consent Form (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT02348853/ICF_000.pdf